CLINICAL TRIAL: NCT00002681
Title: Humanized Anti-Tac Antibody Therapy In Hodgkin's Disease, A Phase Ib/II Trial
Brief Title: Monoclonal Antibody Plus Interleukin-2 in Treating Patients With Leukemia or Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roger Williams Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Richard Junghans, Roger Williams Medical Center
Purpose: Treatment
Other Study IDs: CDR0000064351; BIDMC-92020534; NEDH-92020534; BIDMC-FDR001054; NCI-H95-0732
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Leukemia; Lymphoma
Keywords: recurrent adult Hodgkin lymphoma; recurrent adult acute myeloid leukemia; relapsing chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; atypical chronic myeloid leukemia, BCR-ABL negative
MeSH Terms: conditions — Leukemia; Lymphoma; Hodgkin Disease; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative | interventions — aldesleukin; Daclizumab

INTERVENTIONS:
Biological: aldesleukin
Biological: daclizumab

SUMMARY:
RATIONALE: Monoclonal antibodies can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. Interleukin-2 may stimulate a person's white blood cells to kill leukemia or lymphoma cells. Combining these two therapies may be an effective treatment for leukemia and lymphoma.

PURPOSE: Phase I/II trial to study the effectiveness of monoclonal antibody therapy plus interleukin-2 in treating patients who have leukemia or lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the safety and tolerability of a multidose regimen of humanized anti-Tac monoclonal antibody (HAT) and interleukin-2 (IL-2) in patients with leukemia and lymphoma.
* Describe the pharmacokinetics/pharmacodynamics of HAT and IL-2 in a multidose schedule, including serum half-life of free HAT, area under the curve, and volume of distribution.
* Evaluate the immunogenicity of HAT.
* Identify immunologic parameters that correlate with efficacy.
* Evaluate the preliminary efficacy of HAT in these patients.
* Monitor patients receiving indium-111-labeled HAT for circulating infused antibody for pharmacokinetics, tumor imaging, and bioactivity (binding ability).

OUTLINE: Patients are stratified according to disease (Hodgkin's lymphoma vs acute myelogenous leukemia vs chronic myelogenous leukemia).

Patients receive humanized anti-TAC monoclonal antibody (HAT) IV over 30 minutes on day 1, then IV over 30 minutes every 7 days and interleukin-2 subcutaneously daily. Treatment continues for up to 1 year in the absence of disease progression, unacceptable toxicity, or development of neutralizing antibodies.

Patients are followed weekly for 2 months.

PROJECTED ACCRUAL: A total of 25 patients with Hodgkin's lymphoma and 14 each with AML and CML will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed diagnosis of one of the following malignancies:

  * Hodgkin's lymphoma
  * Acute myelogenous leukemia
  * Chronic myelogenous leukemia
* Failed standard therapy or in chronic phase if on standard therapy
* At least 30% of malignant cells reactive with anti-Tac as determined by immunofluorescence studies

  * All Hodgkin's lymphoma patients eligible due to 100% Tac-positivity of Reed-Sternberg cells
* Measurable disease
* No symptomatic CNS disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* 0-2

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin no greater than 3 times normal
* No significant hepatic disease

Renal:

* Creatinine no greater than 3 times normal
* No significant renal disease

Cardiovascular:

* No significant cardiovascular disease

Pulmonary:

* No significant pulmonary disease

Other:

* No significant endocrine, rheumatologic, or allergic disease
* No HIV-I antibody
* No active disease due to any of the following:
* Cytomegalovirus Herpes simplex virus I/II
* Hepatitis B or C Tuberculosis
* Negative pregnancy test required of fertile women

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior murine anti-Tac monoclonal antibody

Chemotherapy:

* At least 4 weeks since chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* At least 4 weeks since radiotherapy

Surgery:

* Not specified

Other:

* Concurrent treatment allowed for complications of primary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 1995-07; Primary Completion 2003-09 (Actual); Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard P. Junghans, MD, PhD, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States